CLINICAL TRIAL: NCT02880241
Title: An Open Label Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Dose of MMV390048 in Adult Patients With Acute, Uncomplicated Plasmodium Vivax or Falciparum Malaria Monoinfection Over a 35 Day Period
Brief Title: MMV390048 POC in Patients With P. Vivax and P. Falciparum Malaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a Medicines for Malaria Venture (MMV) strategic business decision
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: University of Gondar (Other); Jimma University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_MMV390048_16_02
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — MMV390048

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1A - P. vivax malaria (Experimental): A single oral dose of up to 120mg MMV390048
  Interventions: Drug: MMV390048
- Cohort 1B - P. falciparum malaria (Experimental): A single oral dose of up to 120mg MMV390048
  Interventions: Drug: MMV390048
- Cohort 2A - P. vivax malaria (Experimental): A single oral dose (to be determined) of MMV390048
  Interventions: Drug: MMV390048
- Cohort 2B - P. falciparum malaria (Experimental): A single oral dose (to be determined) of MMV390048
  Interventions: Drug: MMV390048
- Cohort 3A - P. vivax malaria (Experimental): A single oral dose (to be determined) of MMV390048
  Interventions: Drug: MMV390048
- Cohort 3B - P. falciparum malaria (Experimental): A single oral dose (to be determined) of MMV390048
  Interventions: Drug: MMV390048

INTERVENTIONS:
Drug: MMV390048 — Tablets of 20mg each

SUMMARY:
The present proof-of-concept Phase IIa study aims to confirm, in patients, the observed activity of MMV390048 against P. falciparum in pre-clinical models and the human Induced Blood-Stage Malaria (IBSM) challenge model, and to determine the activity against P. vivax malaria in patients, both over 14 and 28 days. Additional aims are to characterise the safety of MMV390048 in patients. Patient safety will be monitored for up to 35 days post-dose including pharmacokinetic assessments. The study will investigate descending single doses of MMV390048 in response to results obtained in the first cohort/dose in each malaria sub-type. The results of this trial will identify active, well-tolerated doses for investigation in combination with a partner drug within a Phase IIb clinical trial.

DETAILED DESCRIPTION:
The present Phase IIa study aims to confirm, in patients, the observed activity of MMV390048 against P. falciparum in pre-clinical models and the human IBSM human challenge model, and to determine the activity against P. vivax malaria in patients, both over 14 and 28 days. Additional aims are to characterise the safety of MMV390048 in patients. Patient safety will be monitored for up to 35 days post-dose including pharmacokinetic assessments. The study will investigate descending single doses of MMV390048 in response to results obtained in the first cohort/dose in each malaria sub type.

The results of this trial will identify active, well tolerated doses for investigation in combination with a partner drug within a Phase IIb clinical trial.

Preclinical studies using SCID mice inoculated with P. falciparum-infected red blood cells link doses and exposures to the efficacy of MMV390048.38 The active dose in the SCID model causing maximum effect (ED90) against the parasites is 1 mg/kg/day. The MPC derived from the SCID data was 39 ng/ml.39 A human dose for the treatment of P. falciparum was sought that could maintain blood concentrations above 39 ng/ml (100 nM) for 8 days. Assuming linear pharmacokinetics and based on observed data from the Phase I exploratory formulation study in human volunteers, a dose of approximately 20 mg would be estimated to achieve the pharmacodynamic target drug concentration in humans based on the preclinical efficacy data generated in the SCID mice model. For new antimalarial drugs the translation of a predicted efficacious dose from the SCID mouse to the human challenge model and in turn to the treatment of acute, uncomplicated P. vivax or P. falciparum is unknown. To minimise the risk to patients and to ensure the highest probability of success, the maximum safe dose (as determined in healthy volunteers) that maintains a toxicokinetic safety margin to the repeat dose studies was selected for the first cohort in this study. This dose is expected to exceed the predicted MPC on Day 8 and provide significant target coverage at the site of action.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 40 kg and 90 kg inclusive
* Presence of P. vivax or P. falciparum monoinfection confirmed by:
* Fever, as defined by axillary temperature ≥37.5°C or oral/rectal/tympanic temperature ≥38°C, or history of fever in the previous 48 hours for P. vivax and 24 hours for P. falciparum and,
* Microscopically confirmed parasite infection: 1,000 to 40,000 asexual parasite count/µL blood
* Written informed consent provided by the patient in accordance with local practice. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations.
* Ability to swallow oral medication
* The patient is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned
* Willing to be hospitalized for at least 72 hours or until malarial parasites are not detected by microscopy on 2 consecutive occasions whichever comes later and return to clinic for all follow-up visits
* Women must be of non-childbearing potential (WNCBP) as per one of the following definitions:
* postmenopausal defined as having age-appropriate, natural (spontaneous) amenorrhea for at least 12 months prior to screening in the absence of an alternative medical cause for the amenorrhea, or
* premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months prior to screening (as determined by subject medical history)
* Sexually active men must agree to comply with strict appropriate contraception rules (barrier contraception, e.g. condom) or complete abstinence when this is in line with the preferred and usual lifestyle of the patient. The contraception coverage in this situation should ensure full elimination of MMV390048, i.e. until 120 days after MMV390048 administration to the enrolled male patient (covering a full sperm cycle of 90 days starting after 5 x t½ of the drug). Abstinent patients must agree to use the above-mentioned contraceptive methods if they start sexual relationships during the study, and to continue these methods until 120 days after study medication.

Exclusion Criteria:

* Patients with signs and symptoms of severe / complicated malaria according to the World Health Organisation Criteria 2012
* Mixed Plasmodium infection
* Vomiting more than three times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment, or diarrhea equivalent to three or more watery stools per day
* Women who are nursing (lactating)
* Presence of other serious or chronic clinical condition requiring hospitalisation
* Severe malnutrition (defined as a body mass index [BMI] of less than 16 kg/m2 as per local guidelines)
* Presence of concurrent febrile illness (e.g. typhoid fever)
* Known history or evidence of clinically significant:
* cardiovascular disease (including arrhythmia, QTcF interval >450 msec, personal or family history of long QT syndrome, PR interval >200msec; any relevant intra-ventricular heart block [QRS >120msec]),
* respiratory conditions (including active tuberculosis),
* history of jaundice or other hepatic dysfunction,
* renal insufficiency,
* gastrointestinal disorder, or any condition that may affect absorption of the study medication (e.g. vomiting or diarrhea),
* immunological disorders (including known pre-existing HIV infection),
* endocrine disorders (including any type of diabetes mellitus whether controlled or not, diabetes insipidus, uncontrolled hypo- or hyperthyroidism, endocrine reproductive disorders not requiring concurrent medication, disorders of adrenal function),
* infectious conditions (other than minor skin or soft tissue infections or confirmed minor lower urinary tract infection),
* malignancy,
* psychiatric or neurological disorders (including a history of convulsions, major head trauma, focal neurological signs, psychosis, bipolar or major depressive disorder), or
* any other disorder or condition that in the opinion of the investigator may render the patient unfit for participation in the trial, may limit his/her ability to provide informed consent, may interfere with protocol adherence or place the patient at increased risk through participation in the study
* Known to have any of the following markers of active hepatitis:
* Hepatitis A IgM (HAV-IgM),
* Hepatitis B surface antigen (HBsAg), or
* Hepatitis C antibody (HCV Ab) and HCV RNA
* Have received any antimalarial treatment (alone or in combination) during the following periods before screening (list of prohibited medication is provided in Appendix 2):
* Piperaquine, mefloquine, naphthoquine or sulphadoxine-pyrimethamine within 6 weeks prior to screening
* Amodiaquine, chloroquine, pyronaridine or tafenoquine within 4 weeks prior to screening
* Any artemisinin derivative (artesunate, artemether, arteether or dihydroartemisinin), quinine, halofantrine, lumefantrine and any other anti-malarial treatment or antibiotic with antimalarial activity (including cotrimoxazole, tetracyclines, quinolones and fluoroquinolones and azithromycin) within 14 days prior to screening
* Any herbal products or traditional medicines during the 7 days prior to screening
* Receipt of an investigational drug within 8 weeks or 5 half-lives (whichever is longer) prior to screening
* Current participation in any other clinical trial
* A history of regular abuse of alcohol, or use of drugs of abuse during the past 6 months, or any clinical signs of substance abuse
* Neutrophil count <1,000/µL
* Elevated liver function tests as follows:
* AST/ALT >2 x the upper limit of normal (ULN), regardless of the level of total bilirubin
* AST/ALT >1.5 and ≤2 x ULN and total bilirubin >ULN
* AST/ALT >ULN and ≤1.5 x ULN
* and total bilirubin >1.5 and ≤2 x ULN,
* and conjugated bilirubin ≥35% of the total bilirubin
* Total bilirubin >2 x ULN, regardless of the level of AST/ALT
* Hb level <8g/dL
* Serum creatinine levels >2 x ULN
* Platelet level <50,000/mm3.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esayas Gudina, MD, Principal Investigator — Jimma University; Mezgebu Silamsaw, MD, Principal Investigator — University of Gondar
Locations (2):
- Ethiopia (2):
  - University of Gondar Hospital/Maksegnit Health Centre, Gonder, Amhara
  - Jimma University Referral Hospital/Agaro District Hospital, Jimma, Oromiya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammed R, Asres MS, Gudina EK, Adissu W, Johnstone H, Marrast AC, Donini C, Duparc S, Yilma D. Efficacy, Safety, Tolerability, and Pharmacokinetics of MMV390048 in Acute Uncomplicated Malaria. Am J Trop Med Hyg. 2022 Dec 5;108(1):81-84. doi: 10.4269/ajtmh.22-0567. Print 2023 Jan 11. PMID 36509063

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1A - P. Vivax Malaria | Cohort 1B - P. Falciparum Malaria | Cohort 2A - P. Vivax Malaria | Cohort 2B - P. Falciparum Malaria | Cohort 3A - P. Vivax Malaria | Cohort 3B - P. Falciparum Malaria
Started | 8 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated)
Completed | 7 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated) | 0 (Study terminated)
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated prior to completion of Cohort 1A - P. vivax, and recruitment of any of Cohort 1B -P. falciparum participants. There were no participants in Cohort 1 B-P. falciparum to contribute to the Primary endpoint data.
  Cohort 2 A - P. vivax, Cohort 2B - P. falciparum, Cohort 3A - P. vivax and Cohort 3B - P falciparum malaria did not enrol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A - P. Vivax Malaria | Cohort 1B - P. Falciparum Malaria | Cohort 2A - P. Vivax Malaria | Cohort 2B - P. Falciparum Malaria | Cohort 3A - P. Vivax Malaria | Cohort 3B - P. Falciparum Malaria | Total
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  |  |  | 0
  Between 18 and 65 years | 8 |  |  |  |  |  | 8
  >=65 years | 0 |  |  |  |  |  | 0
Age, Continuous [Median (Full Range); unit: Years] | 24.5 [20 to 50] |  |  |  |  |  | 24.5 [20 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  |  |  |  | 0
  Male | 8 |  |  |  |  |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  |  |  | 0
  Not Hispanic or Latino | 8 |  |  |  |  |  | 8
  Unknown or Not Reported | 0 |  |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  |  | 0
  Asian | 0 |  |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  |  | 0
  Black or African American | 8 |  |  |  |  |  | 8
  White | 0 |  |  |  |  |  | 0
  More than one race | 0 |  |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  Ethiopia | 8 |  |  |  |  |  | 8
Pre-dose asexual parasite count [Mean (Standard Deviation); unit: asexual parasite/μL] — Pre-dose asexual parasite count for P. vivax determined by microscopy
  asexual parasite/μL | 6405.5 (6766.6) |  |  |  |  |  | 6405.5 (6766.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.1 (1.20) |  |  |  |  |  | 18.1 (1.20)
Pre-dose gametocyte count [Mean (Standard Deviation); unit: gametocyte/μL] — Pre-dose gametocyte count for P. vivax determined by microscopy.
  gametocyte/μL | 268.5 (355.2) |  |  |  |  |  | 268.5 (355.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Crude Adequate Clinical and Parasitological Response (ACPR) for P. Vivax
Description: The absence of parasitaemia (thick smear) on Day 14, irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure. Parasitaemia was defined as a P. vivax asexual forms count >0
Time Frame: On Day 14 post-dose
Population: All enrolled participants who received any amount of study medication.
Measure: Number; unit: participants
Arm/Group | Cohort 1B - P. Falciparum Malaria | Cohort 1A - P. Vivax Malaria | Cohort 2A - P. Vivax Malaria | Cohort 2B - P. Falciparum Malaria | Cohort 3A - P. Vivax Malaria | Cohort 3B - P. Falciparum Malaria
Number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0
participants |  | 8 |  |  |  |

2. Primary Outcome: For P. Falciparum: PCR-adjusted Crude Adequate Clinical and Parasitological Response (ACPR)
Description: Number of participants meeting PCR-adjusted Crude Adequate Clinical and Parasitological Response (ACPR)
Time Frame: On Day 14 post-dose
Population: Cohort 1B - P falciparum malaria did not enroll participants.
Arm/Group | Cohort 1A - P. Vivax Malaria | Cohort 1B - P. Falciparum Malaria | Cohort 2A - P. Vivax Malaria | Cohort 2B - P. Falciparum Malaria | Cohort 3A - P. Vivax Malaria | Cohort 3B - P. Falciparum Malaria
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From IMP administration (Day 0) to End of Study (Day 35)
Description: SAEs will be recorded from the time of screening until the end of study, and additionally until 30 days after completion of the study should the Investigator be made aware of such an event.
Arm/Group | Cohort 1B - P. Falciparum Malaria | Cohort 1A - P. Vivax Malaria | Cohort 2A - P. Vivax Malaria | Cohort 2B - P. Falciparum Malaria | Cohort 3A - P. Vivax Malaria | Cohort 3B - P. Falciparum Malaria
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/8 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/8 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 8/8 | 0/0 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1B - P. Falciparum Malaria (N=0) | Cohort 1A - P. Vivax Malaria (N=8) | Cohort 2A - P. Vivax Malaria (N=0) | Cohort 2B - P. Falciparum Malaria (N=0) | Cohort 3A - P. Vivax Malaria (N=0) | Cohort 3B - P. Falciparum Malaria (N=0)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Ascariasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hookworm infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
P.falciparum infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02880241/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02880241/SAP_001.pdf